CLINICAL TRIAL: NCT03524846
Title: Effect of Ascorbic Acid Administration on Restenosis of Dysfunctional Hemodialysis Vascular
Brief Title: Ascorbic Acid on Restenosis of Dysfunctional Hemodialysis Vascular Access
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Principal Investigator, IRB of NTUH Hsin-Chu Branch, Secretary In Medical Affairs/Director of Nephrology, National Taiwan University Hospital Hsin-Chu Branch
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99G002
Record Dates: First submitted 2018-04-30; First posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Hemodialysis Access Failure
Keywords: Ascorbic acid; hemodialysis vascular access; restenosis
MeSH Terms: interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: This was a prospective randomized, single-blind, placebo-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ascorbic acid 300 mg (Active Comparator): Ascorbic acid 300 mg was administered intravenously for 5 minutes after each dialysis session, three times per week for 12 weeks.
  Interventions: Drug: Ascorbic Acid 300 MG
- Ascorbic acid 600 mg (Active Comparator): Ascorbic acid 600 mg was administered intravenously for 5 minutes after each dialysis session, three times per week for 12 weeks.
  Interventions: Drug: Ascorbic Acid 600 MG
- Placebo (Placebo Comparator): Normal saline was administered intravenously for 5 minutes after each dialysis session, three times per week for 12 weeks.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ascorbic Acid 300 MG — Ascorbic acid 300 mg was administered intravenously for 5 minutes after each dialysis session, three times per week for 12 weeks.
  Other Names: Vitamin C
  Arms: Ascorbic acid 300 mg
Drug: Ascorbic Acid 600 MG — Ascorbic acid 600 mg was administered intravenously for 5 minutes after each dialysis session, three times per week for 12 weeks.
  Other Names: Vitamin C
  Arms: Ascorbic acid 600 mg
Drug: Normal saline — Normal saline was administered intravenously for 5 minutes after each dialysis session, three times per week for 12 weeks.
  Arms: Placebo

SUMMARY:
To investigate the effect of ascorbic acid on angiographic restenosis after percutaneous transluminal angioplasty (PTA) for dysfunctional dialysis vascular access.

DETAILED DESCRIPTION:
Vascular access dysfunction is the leading cause of treatment insufficiency or interruption among hemodialysis (HD) patients, and it is responsible for a large portion of the cost of any end-stage renal disease (ESRD) program. Intimal hyperplasia at the venous segment of vascular access is the characteristic lesion, which leads to dysfunction or failure of both arteriovenous fistulas (AVF) and prosthetic grafts (AVG). Although percutaneous transluminal angioplasty (PTA) is effective in treating these stenotic lesions, the effect seems not permanent and restenosis after PTA remains a major problem. A number of studies have examined the clinical, anatomical, and technical factors for restenosis, the causes of restenosis are still not fully understood.This highlights a possible role of non-traditional risk factors to explain the high restenosis rate at the venous segment of vascular access, which includes oxidative stress, inflammation, and endothelial dysfunction.

Ascorbic acid (vitamin C) is a potent antioxidant used for a long time. Hemodialysis patients had been shown to be deficient in antioxidant defense, which resulted in increasing requirement of ascorbic acid supplement. Currently, intravenous 300-mg ascorbic acid supplementation three times a week after hemodialysis had been used to overcome erythropoietin resistance in patients with iron deficiency. Theoretically, ascorbic acid scavenges reactive oxygen species and reactive nitrogen species and may thereby prevent oxidative injuries. Investigators reported that administration of high dose ascorbic acid could prevent lipid peroxidation and oxidative DNA damage in patients with ESRD.

In this study, the investigators investigated whether ascorbic acid could decrease venous restenosis after PTA for dysfunctional hemodialysis vascular access.

ELIGIBILITY:
Inclusion Criteria:

* clinical signs, i.e., decreased thrill, development of collateral veins, limb swelling, and prolonged bleeding from puncture sites, suggesting vascular access dysfunction
* reduction of flow rate more than 25% from baseline
* total access blood flow rate less than 500 mL/min by ultrasound dilution method
* increased venous pressure during dialysis, as dynamic venous pressure exceeding threshold levels of 150 mmHg in AVF and 160 mmHg in AVG, respectively, under dialysis blood flow 250 ml/min for three consecutive times

Exclusion Criteria:

* hospitalized for infection, heart failure, or acute coronary syndrome in recent 3 months
* unable to comply with follow-up visits
* already under ascorbic acid or other antioxidant supplements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
the extent of restenosis after angioplasty | 12 weeks
  the extent of restenosis defined by the late loss of minimal vessel diameter and late loss of percentage stenosis at follow-up angiograms

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Cheng Wu, M.D., Study Director — Associate professor of Medicine, National Taiwan University, College of Medicine, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tomoda H, Yoshitake M, Morimoto K, Aoki N. Possible prevention of postangioplasty restenosis by ascorbic acid. Am J Cardiol. 1996 Dec 1;78(11):1284-6. doi: 10.1016/s0002-9149(96)00613-3. PMID 8960592
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Yang CW, Wu CC, Luo CM, Chuang SY, Chen CH, Shen YF, Tarng DC. A randomized feasibility study of the effect of ascorbic acid on post-angioplasty restenosis of hemodialysis vascular access (NCT03524846). Sci Rep. 2019 Jul 31;9(1):11095. doi: 10.1038/s41598-019-47583-w. PMID 31366980